CLINICAL TRIAL: NCT00988858
Title: A Phase 2 Study to Evaluate LY2603618 in Combination With Pemetrexed in Patients With Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: A Study of Advanced or Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12092; I2I-MC-JMMD (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — LY2603618; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2603618 and Pemetrexed (Experimental)
  Interventions: Drug: LY2603618; Drug: Pemetrexed

INTERVENTIONS:
Drug: LY2603618 — 150 milligram per square meter (mg/m^2) intravenously on Day 2 of each 21 day cycle repeating every 21 days for a minimum of 2 cycles continuing until disease progression
Drug: Pemetrexed — 500 mg/m^2 intravenously on Day 1 of each 21 Day cycle repeating every 21 days for a minimum of 2 cycles or until disease progression
  Other Names: Alimta; LY231514

SUMMARY:
The primary purpose of this study is to evaluate the efficacy and safety of LY2603618 in combination with pemetrexed and any side effects that might be associated with it along with determining the effects of LY2603618 in combination with pemetrexed in participants with advanced or metastatic Non-small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Must agree to have a tumor biopsy at screening
* Must have a diagnosis of advanced or metastatic non-squamous non-small cell lung cancer that has progressed after certain prior treatment
* Must be available for the duration of the study and willing to follow the study procedures
* If participant is a woman that is capable of having children, must have a negative pregnancy test within 7 days of taking first dose of study drug
* Must have discontinued radiation therapy at least 4 weeks before entering this study

Exclusion Criteria:

* Must not have taken an unapproved drug as treatment for any indication within the last 28 days before starting study treatment.
* Must not be pregnant or lactating, are considering becoming pregnant, or are considering fathering a child. Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial until the participant's physician considers it safe to become pregnant or father a child.
* Must not have known positive test in human immunodeficiency virus (HIV), hepatitis B surface antigen (HBSAg), or hepatitis C antibodies (HCAb).
* Must not have previously participated in a study involving LY2603618
* Must not have previously taken pemetrexed for cancer
* Must not have a known allergy to LY2603618 or pemetrexed
* Must not currently have an infection that may affect participant's ability to tolerate the therapy
* Must not have a serious medical condition or disorder that would make it unsafe for you to participate in the study such as uncontrolled diabetes or chest pain due to heart disease
* If taking certain medications called non-steroidal anti-inflammatory drugs (NSAIDS), such as ibuprofen, must be able to stop taking these medications according to certain guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-11; Primary Completion 2012-07 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kettering, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tyler, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yakima, Washington
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orbassano, Italy
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea
- Taiwan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Scagliotti G, Kang JH, Smith D, Rosenberg R, Park K, Kim SW, Su WC, Boyd TE, Richards DA, Novello S, Hynes SM, Myrand SP, Lin J, Smyth EN, Wijayawardana S, Lin AB, Pinder-Schenck M. Phase II evaluation of LY2603618, a first-generation CHK1 inhibitor, in combination with pemetrexed in patients with advanced or metastatic non-small cell lung cancer. Invest New Drugs. 2016 Oct;34(5):625-35. doi: 10.1007/s10637-016-0368-1. Epub 2016 Jun 27. PMID 27350064

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants that had progressive disease were completers.
Groups:
- LY2603618 and Pemetrexed: LY2603618: 150 milligram per square meter mg/m^2 intravenously on Day 2 of each 21 day cycle repeating every 21 days for a minimum of 2 cycles or until disease progression
  Pemetrexed: 500mg/m^2 intravenously on Day 1 of each 21 Day cycle repeating every 21 days for a minimum of 2 cycles or until disease progression
Period: Overall Study
Arm/Group | LY2603618 and Pemetrexed
Started | 55
Completed | 45
Not Completed | 10
Not completed — Adverse Event | 7
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Sponsor Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- LY2603618 and Pemetrexed: LY2603618: 150 mg/m2 intravenously on Day 2 of each 21 day cycle repeating every 21 days for a minimum of 2 cycles continuing until disease progression
  Pemetrexed: 500mg/m2 intravenously on Day 1 of each 21 Day cycle repeating every 21 days for a minimum of 2 cycles or until disease progression
Arm/Group | LY2603618 and Pemetrexed
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
  Taiwan | 5
  Korea, Republic of | 14
  Italy | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Tumor Response - Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) [Overall Response Rate (ORR)]
Description: Overall response rate is the best response of complete response (CR) or partial response (PR) as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of not-target lesions or appearance of new lesions. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants with at least 1 measurable lesion, multiplied by 100.
Time Frame: Baseline until Progressive Disease or Study Discontinuation (Up to 23 Months)
Population: All randomized participants who received at least 1 dose of drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LY2603618 and Pemetrexed
Number analyzed (Participants) | 55
percentage of participants | 9.1 [3.7 to 18.2]

2. Secondary Outcome: Percentage of Participants Who Achieved a Best Response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) (Clinical Benefit Rate)
Description: Clinical benefit rate is the best response CR, PR, or stable disease (SD) as classified by the investigators according to the RECIST v1.1. CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of not-target lesions or appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameter since treatment started. Clinical benefit rate is calculated as a total number of participants with CR, PR, or SD divided by the total number of participants with at least 1 measurable lesion, multiplied by 100.
Time Frame: Baseline until Progressive Disease or Study Discontinuation (Up to 23 Months)
Population: All randomized participants who received at least 1 dose of drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | LY2603618 and Pemetrexed
Number analyzed (Participants) | 55
percentage of participants | 45.5 [33.9 to 57.4]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) time was defined as the time from the date of randomization to the first date of progressive disease (symptomatic or objective) or death due to any cause, whichever occurred first. For participants who were not known to have died or progressed as of the data-inclusion cutoff date, PFS time was censored at the date of the last objective progression-free disease assessment prior to the date of any subsequent systematic anticancer therapy. PFS was summarized using Kaplan-Meier estimates.
Time Frame: Baseline to Progressive Disease or Death Due to Any Cause (Up to 27.1 Months)
Population: All randomized participants who received at least 1 dose of drug. 9 participants were censored.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LY2603618 and Pemetrexed
Number analyzed (Participants) | 55
months | 2.3 [1.4 to 3.3]

4. Secondary Outcome: Duration of Response
Description: Duration of Response is defined as the time from the first observation of CR or PR to the first observation of progressive disease (PD) or death from any cause. A response is defined as a confirmed objective status of CR or PR. For participants who are not known to have died as of the data inclusion cut-off date and who do not have PD, the duration will be censored at the date of the last objective progression free disease assessment prior to the date of any subsequent anticancer therapy.
Time Frame: First Observation of CR or PR until Progressive Disease or Death Due to Any Cause (Up to 23 Months)
Population: All randomized participants who received at least 1 dose of drug with Best Overall Response of Complete Response or Partial Response.5 participants were censored.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LY2603618 and Pemetrexed
Number analyzed (Participants) | 55
months | 8.7 [7.0 to NA] — Upper limit is not estimable based on sample size.

5. Secondary Outcome: Change in Symptom Burden Scores of Lung Cancer Symptom Scale (LCSS)
Description: The LCSS participants scale is a 9-item questionnaire. Six questions are symptom-specific measures for lung cancer (appetite, fatigue, cough, dyspnea, hemoptysis and pain), and 3 summation items describe total symptomatic distress, activity status, and overall quality of life. Participant responses were measured using visual analogue scales (VAS) with 100-milliliter (mm) lines. Scores range from 0 (for best outcome) to 100 (for worst outcome). The Average Symptom Burden Index (ASBI) was calculated as the mean of 6 symptom-specific questions from the LCSS.
Time Frame: Baseline until End of Study (Up to 27.1 Months)
Population: The LCSS evaluable population consisted of all enrolled participants who had a baseline LCSS measurement and at least 1 post-baseline measurement. The population was evaluated for changes in the ASBI (improved, stable, worsened), with improvement/worsening based on trends seen in sets of consecutive ASBI assessments with respect to baseline ASBI.
Measure: Number; unit: participants
Arm/Group | LY2603618 and Pemetrexed
Number analyzed (Participants) | 46
participants
  Improved | 12
  Worsened | 6
  Stable | 18
  Unknown | 10

6. Secondary Outcome: Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) of LY2603618
Time Frame: Day 2 and Day 3 of Cycle 1 and Cycle 2: Prior to End of Infusion (EOI); EOI + 1-2 hr; EOI + 4-6 hr; EOI + 20-28 hr; anytime on Day 8 of Cycle 1 and Cycle 2
Population: All randomized participants who received at least 1 dose of drug and evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | LY2603618 and Pemetrexed
Number analyzed (Participants) | 48
nanogram per milliliter (ng/mL)
  Day 2/Cycle 1 (n=41) | 3430 (50)
  Day 2/Cycle 2 (n=48) | 3560 (40)

7. Secondary Outcome: PK: Maximum Plasma Concentration (Cmax) of Pemetrexed
Time Frame: Day 1 and Day 2 of Cycle 1 and Cycle 2: Prior to End of Infusion (EOI); EOI + 1-2 hour (hr); EOI + 4-6- hr; EOI + 20-28 hr
Population: All randomized participants who received at least 1 dose of drug and evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | LY2603618 and Pemetrexed
Number analyzed (Participants) | 43
microgram per milliliter (μg/mL)
  Day 1/Cycle 1 (n=40) | 102 (50)
  Day 1/Cycle 2 (n=43) | 96.8 (42)

8. Secondary Outcome: PK: Area Under the Plasma Concentration vs. Time Curve From Time Zero to Infinity [AUC(0-∞)] of LY2603618
Time Frame: as for outcome 6
Population: All randomized participants who received at least 1 dose of drug and had evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | LY2603618 and Pemetrexed
Number analyzed (Participants) | 48
nanograms*hour per milliliter (ng*h/mL)
  Day 2/Cycle 1 (n=41) | 38000 (85)
  Day 2/Cycle 2 (n=48) | 41500 (88)

9. Secondary Outcome: PK: Area Under the Plasma Concentration vs. Time Curve From Time Zero to Infinity [AUC(0-∞)] of Pemetrexed
Time Frame: as for outcome 7
Population: All randomized participants who received at least 1 dose of drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (µg*hr/mL)
Arm/Group | LY2603618 and Pemetrexed
Number analyzed (Participants) | 43
microgram*hour per milliliter (µg*hr/mL)
  Day 1/Cycle 1(n=40) | 193 (31)
  Day 1/Cycle 2(n=43) | 202 (33)

ADVERSE EVENTS:
Arm/Group | LY2603618 and Pemetrexed
Serious Adverse Events (participants affected / at risk) | 16/55
Other Adverse Events (participants affected / at risk) | 51/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2603618 and Pemetrexed (N=55)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2603618 and Pemetrexed (N=55)
Anaemia (Blood and lymphatic system disorders) | 10 (12)
Leukopenia (Blood and lymphatic system disorders) | 8 (13)
Neutropenia (Blood and lymphatic system disorders) | 15 (35)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (6)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 11 (15)
Diarrhoea (Gastrointestinal disorders) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 18 (28)
Stomatitis (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 12 (12)
Face oedema (General disorders) | 4 (4)
Fatigue (General disorders) | 20 (27)
Pyrexia (General disorders) | 5 (5)
Herpes zoster (Infections and infestations) | 3 (3)
Alanine aminotransferase increased (Investigations) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 4 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Flushing (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days